CLINICAL TRIAL: NCT05767281
Title: Comparative Evaluation of Comprehensive Programs for the Prevention of Dental Diseases for the Children's Population of Chapaevsk
Brief Title: Comparative Evaluation of Dental Disease Prevention Programs
Status: Active, not recruiting | Type: Observational
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 13
Record Dates: First submitted 2023-02-05; First posted 2023-03-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Carious and Non-carious Lesions of the Teeth
Keywords: ecology;; children caries;; periodontal diseases;; epidemiology;; prevalence of caries;; intensity of caries.
MeSH Terms: conditions — Periodontal Diseases | interventions — National Program of Cancer Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Urine and oral fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Children 3 years old: Epidemiological examination of children according to the WHO 2013 methodology, including only an examination of the oral cavity.
  Interventions: Behavioral: prevention program
- Children 5-6 years old: Epidemiological examination of children according to the WHO 2013 methodology, including only an examination of the oral cavity.
  Interventions: Behavioral: prevention program
- Children 7 years old: Epidemiological survey of adolescents according to the WHO 2013 methodology, including only an examination of the oral cavity.
  Interventions: Behavioral: prevention program
- Children 12 years old: Epidemiological survey of adolescents according to the WHO 2013 methodology, including an examination of the oral cavity and a questionnaire.
  Interventions: Behavioral: prevention program
- Teenagers 15 years old: Epidemiological survey of adolescents according to the WHO 2013 methodology, including an examination of the oral cavity and a questionnaire.
  Interventions: Behavioral: prevention program
- Teenagers 18 years old: Epidemiological survey of adolescents according to the WHO 2013 methodology, including an examination of the oral cavity and a questionnaire.
  Interventions: Behavioral: prevention program

INTERVENTIONS:
Behavioral: prevention program — introduction of the developed comprehensive prevention program among the child population with the participation of primary health care personnel, which will improve not only the dental health of children, their quality of life, but will also help reduce foci of chronic oral sepsis.

SUMMARY:
Relevance. The dental health of the Chapaevsk children's population and the risk factors for dental caries and periodontal disease were well studied in 1995-2009. But pilot epidemiological studies conducted in 2018 by employees of the Department of Pediatric Dentistry and Orthodontics showed that despite the improvement in the environmental situation as a result of large-scale state measures of the city's environmental rehabilitation program, the prevalence and intensity of dental caries increased against the background of improved somatic health indicators. In addition, the "K" component (untreated caries) prevails in the structure of the KPU, which indicates gaps in the organization of dental care.

At present, the development and implementation of a comprehensive program for the prevention of dental diseases, based on an analysis of the situation and aimed at strengthening the health and improving the quality of life of children in Chapaevsk, remains an extremely urgent problem. Such a program can be used for implementation in other regions with the adaptation of measurable prevention targets.

Scientific novelty of the research. Identification of risk factors affecting children's dental health, especially regarding the safety of using fluoride to prevent dental caries Development of a comprehensive program for the prevention of the child population, taking into account the analysis of the situation in dentistry in Chapaevsk, with the participation of primary health care personnel, caregivers and families.

The practical significance of the study involves the introduction of a developed comprehensive prevention program among the child population, based on interdisciplinary interaction at the level of primary health care and interdepartmental interaction with the teaching staff of preschool educational institutions and schools.

DETAILED DESCRIPTION:
Purpose of the study. Development of a comprehensive program for the prevention of dental caries, periodontal disease based on an analysis of the situation in dentistry.

Research objectives:

1. To study the prevalence and intensity of major dental diseases from 1995 to 2023 according to the WHO methodology (2013);
2. To study the behavioral risk factors for dental diseases in the child population of Chapaevsk according to the WHO methodology (2013);
3. To study the concentration of fluorine ion in the drinking water of municipal water supply and its other sources (bottled water, street vending machines for drinking water, filtered water, etc.);
4. To study the awareness of the population, parents, primary health care personnel, educators, teachers about the risk factors for chronic non-communicable diseases (arterial hypertension, cardiovascular diseases, diabetes mellitus, etc.) and their prevention;
5. To study the features of urinary fluoride excretion in preschool children in order to justify the safety of using fluorides to prevent caries;
6. Conduct an analysis of the situation in dentistry and develop a comprehensive program for the prevention of dental morbidity for the child population;
7. To study in a pilot project the effectiveness of the developed program for the prevention of major dental diseases.

Materials and research methods.

1. Epidemiological studies according to WHO (2013) - 1000 people (3, 5-6, 7 years old, 12, 15, 18 years old) with the WHO questionnaire (parents of children aged 3, 5-6, 7 years and children 12, 15 , 18 years old (1000 people)).
2. Determination of fluorides in public water supply, individual households, bottled water and urine using an F-selective electrode (Mettler Toledo).
3. Determination of F ions before filtration and after filtration of water using household filters.
4. Marketing studies of hygiene products (toothpastes, additional oral hygiene products), in pharmaceutical institutions, markets and markets)
5. Studying the effectiveness of the implemented prevention program by blind control after 3 months, 6 months, 1 year, 1.5 years, 2 years.
6. Statistical analysis of the effectiveness of the prevention program in the pilot project.

Scientific novelty.

* risk factors affecting the dental health of children will be identified;
* a comprehensive program for the prevention of the child population will be developed, taking into account the analysis of the situation in dentistry;
* the need and safety of the use of fluorides for the prevention of dental caries will be justified (based on the study of the proportion of fluorides excreted by the kidneys and the analysis of the intensity of dental caries.

Practical significance.

1. During the study, the timing of the eruption of permanent teeth will be established;
2. Recommendations will be developed to improve the quality and accessibility of dental care;
3. The importance of monitoring fluoride in drinking water and the daily total intake of fluoride in the body of children will be proved by studying the proportion of fluoride excreted by the kidneys to justify safety;
4. The introduction of the developed prevention program will improve the dental health of children;
5. The need for interdisciplinary and interdepartmental interaction to improve the dental health of children will be substantiated.

ELIGIBILITY:
Inclusion Criteria:

* The main age groups of the WHO survey (2013)

Exclusion Criteria:

-

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Dental examination of children will be carried out in the conditions of school educational institutions after obtaining voluntary informed consent for dental examination from the administration and legal representatives of students.
  Examination of children will be carried out directly in the classroom using sterile sets of dental instruments (dental and periodontal probes, dental mirrors).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Index of DMF | 5 minutes
  The decay-missing-filled (DMF) index or decayed, missing, and filled teeth (DMFT) index is one of the most common methods in oral epidemiology for assessing dental caries prevalence as well as dental treatment needs among populations. This index is based on in-field clinical examination of individuals by using a probe, mirror and cotton rolls, and simply counts the number of decayed, missing (due to caries only) and restored teeth. Statistics are available per populations according to age.

CONTACTS AND LOCATIONS:
Locations (1):
- Liliya, Samara, Russia